CLINICAL TRIAL: NCT05739565
Title: Title Impact of a Physical Activity Intervention With Motivational Support From Peers for Prostate Cancer Patients - ACTI-PAIR 2 Multicenter, Randomized Stepped-wedge Study
Brief Title: Impact of a Physical Activity Intervention With Motivational Support From Peers for Prostate Cancer Patients
Acronym: ACTI-PAIR2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: Sport Health Center of Auvergne-Rhône Alpes (Unknown); INSERM, SAINBIOSE U1059 (Unknown); Institut National de la Santé Et de la Recherche Médicale, France (Other Government); INSERM ECEVE 1123 (Unknown); Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 20PH286; 2022-A01094-39 (Other: ANSM)
Record Dates: First submitted 2023-01-26; First posted 2023-02-22 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Prostate Cancer
Keywords: Physical activity; prostate cancer; interventional research
MeSH Terms: conditions — Prostatic Neoplasms; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acti-Pair program (Experimental): * Motivational support by the peer (a patient with the same pathology who meets the WHO recommendations for physical activity), who will provide motivational follow-up
  * The implementation of a personalized and realistic physical activity project for the patient via the physical activity support systems (sport health centers)
  * Support from health professionals (GP) via the prescription of physical activity and from adapted physical activity (APA) professionals
  Interventions: Behavioral: Acti-Pair program
- Usual care (No Intervention): The control group will be made up of patients followed up for prostate cancer and benefiting from usual care which consists of giving advice and recommendations for physical activity in consultation, aiming to make patients more active in their daily lives (=usual practice, physical activity to be carried out independently, at home).

INTERVENTIONS:
Behavioral: Acti-Pair program — Motivational support by the peer (a patient with the same pathology who meets the WHO recommendations for physical activity), who will provide motivational follow-up
  * The implementation of a personalized and realistic physical activity project for the patient via the physical activity support systems (sport health centers)
  * Support from health professionals (GP) via the prescription of physical activity and from adapted physical activity (APA) professionals
  Arms: Acti-Pair program

SUMMARY:
Despite the recognized benefits of physical activity in tertiary prevention, 60-70% of prostate cancer patients are insufficiently active.

Yet 150 minutes of brisk walking per week (new WHO recommendations) is associated with a 29% reduction in cancer mortality and a 57% reduction in recurrence.

Increasing patients' adherence to regular physical activity appears to be a new challenge for personalized cancer care.

Personalized physical activity programmes (1) at home, (2) supported by health professionals, or (3) by peers have shown the effectiveness of regular physical activity.

However, these interventions last less than 6 months and do not allow for long-term sustainability of physical activity.

This study proposes to combine 3 interventions, which aim to initiate and maintain regular physical activity in prostate cancer patients:

* 1-The realization of a personalized and realistic physical activity project via physical activity support devices (sport health centers)
* 2-Coaching by a peer (a patient with the same disease who has reached the WHO recommendations for physical activity), who will provide motivational follow-up
* 3-Support by health professionals (attending physician) through the prescription of physical activity.

The feasibility of ACTI-PAIR program has been demonstrated, the investigators now wish to evaluate it effectiveness.

ELIGIBILITY:
Inclusion Criteria:

Patients:

* Age ≥ 18 years
* Diagnosed with prostate cancer for at least 1 year
* PA practice < 150 minutes per week (considered inactive according to WHO)
* Affiliated or entitled to a social security scheme
* Having received informed information about the study and having co-signed, with the investigator, a consent to participate in the study

Exclusion Criteria:

For patients:

* Undergoing treatment (except hormone therapy)
* Significant comorbidities contraindicating the practice of physical activity: associated cardiac pathologies, respiratory pathologies, disabling joint pathologies
* Deprived of liberty or under guardianship

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 850 (Estimated)
Dates: Start 2023-04-25 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
Objective measurement of physical activity (in MET-hr/week, Metabolic Equivalent of Task (MET), measures the intensity of physical activity) | Month: 12
  via actimetry (Actigraph GT9x, Pensacola, Florida, USA) 12 months (+/- 1 month) after the patient's inclusion in the Acti-Pair program

SECONDARY OUTCOMES:
Objective measurement of physical activity (in MET-hr/week, Metabolic Equivalent of Task (MET), measures intensity of physical activity) | Inclusion, 3, 6 and 12 months
  via actimetry (Actigraph GT9x, Pensacola, Florida, USA) (at 3 and 6 months).
Objective measure of physical inactivity (in h/d) | Inclusion, 3, 6 and 12 months
  via actimetry (Actigraph GT9x, Pensacola, Florida, USA)
Subjective measurement of physical activity (in Metabolic equivalent of task-h/week) and sedentary time (h/d) | Inclusion, 3, 6 and 12 months
  Via the e-Adult Physical Activity Questionnaire (e-APAQ, EA SNA-EPIS, University of Jean Monnet, Saint-Etienne, France) e-Adult Physical Activity Questionnaire (e-APAQ) assesses the 5 categories of physical activity (work, travel, daily life, leisure and sport) and daily life, leisure and sport). The minimum value is 1 and the maximum value is 300. More the physical activity score is high, more the patient is active. This questionnaire authenticates the periods of sedentarity (at work, during travel and daily life, leisure and sport). The minimum value is 1 and the maximum value is 24. More the sedentarity score is high, more the patient is sedentary.
Measurement of physical capacity: walking distance (meters) | Inclusion, 3, 6 and 12 months
  via the 6-minute walk test (6MWT).
Measurement of muscle strength: biceps muscle strength (kg) | Inclusion, 3, 6 and 12 months
  via the handgrip (JAMAR Hand Dynamometer, Nottingham, UK).
Level of fatigue assessed by measuring heart rate variability (SDNN and RMSSD in ms) | Inclusion, 3, 6 and 12 months
  via heart rate monitor connected to an actimeter (Actigraph GT3x, Pensacola, Florida, USA) for 24 hours
Level of fatigue | Inclusion, 3, 6 and 12 months
  via the FACIT-F questionnaire (Functional Assessment of Chronic Illness Therapy - Fatigue Scale). This questionnaire asseses fatigue and it impacts. The score range is 0 to 160. More the score is higher, more the fatigue is high.
Health-related quality of life | Inclusion, 3, 6 and 12 months
  via the EuroQol-5D questionnaire (EQ-5D-5L). The score range is -0.148 to 0.949. Mre the score is high, more the quality of life is good.
Adoption of Acti-Pair program by physicians | through end of inclusion, an average of 30 months
  Number of physicians including patients
Adoption of Acti-Pair program by peers | through end of inclusion, an average of 30 months
  Number of peers recruited
Adoption of Acti-Pair program by Adapted Physical Activity (APA) professionals | through study completion, an average of 42 Months
  Number of patients followed by APA professionals
Time dedicated by peers, Adapted Physical Activity (APA) professionals and health professionals to the Acti-Pair program | through study completion, an average of 42 Months
  Number of hours spend to follow-up patient specifically for the Acti-Pair program by peers, Adapted Physical Activity (APA) professionals and health professionals
Assessment of the context:factors favoring and hindering implementation, achievement, adaptation and sustainability of the programme ; compliance with the programme ; social representations | Before and after the implementation of the intervention
  Semi-structured interviews
Percentage of adherence to the intervention | 12 months
  via the number of patients continuing the programme 12 months after initiation
Motivation to engage in physical activity for patients and peers | Inclusion, 3, 6 and 12 months
  via the behavioural regulation in exercise questionnaire (BREQ-2). This questionnaire consists of 19 items includes 6 sub-scores of motivations : introjected regulation (3 items), external regulation (4 items), intrinsic regulation (4 items), integrated regulation, amotivation (4 items) and identified regulation (4 items) on a scale from 1 (Not at all true for me) to 5 (Absolutely true for me).
Alliance between the patient and the peer | 12 months
  via the Working Alliance Inventory - short version (WAI-SR). This questionnaire measures three dimensions: bonding (development of a positive interpersonal attachment between the patient and the peer including mutual trust and respect), tasks (each partner's perception of the appropriateness and effectiveness of the care tasks, as well as tasks, as well as shared responsibility for their execution) and goals (understanding, validation and acceptance by both partners of the objectives of change in physical activity management).
  Patients rate items on a 5-point Likert scale anchored at each end with 'rarely or never' (1) and 'always' (5). The Goal, Task and Bond domains each have scores ranging from 5 to 20. Higher scores indicate a better therapeutic alliance.
Patients, peers and professionals satisfaction | 12 months
  Via a satisfaction questionnaire constructed for the Acti-Pair programme. The proposed responses are a likert scale ranging from Strongly Agree to Strongly Disagree. Each item will be described with a percentage of Likert scale for each response. More participants will fill out they have been strongly agree, more they will be satisfied.This questionnaire does not have a score.
Cost per quality adjusted life year (QALY) gained through the intervention (quality adjusted life year) | 12 months
  Quality of life data will be collected (e.g. quality of life using the EQ-5D-5L questionnaire, Appendix 3), transformed into utilities to calculate quality adjusted life year (QALY), and the number of patients continuing physical activity at 12 months. Cost data will be collected throughout the study, in each of the 8 departments involved. The analysis will be carried out from the payer's (health insurance) perspective. The time horizon will be that of the study (12 months), and therefore in accordance with French guidelines (HAS), no discount rate will be applied
Cost per patient continuing physical activity at 12 months through the intervention | 12 months
  The costs will include : - direct medical costs : health professionals consultations, peer-to-peer, patient sessions with APA professionals - indirect costs of implementing the intervention: training, facility rental operating costs, investment in small equipment

CONTACTS AND LOCATIONS:
Overall Officials: David HUPIN, MD PhD, Principal Investigator — CHU de Saint-Etienne
Locations (25):
- France (25):
  - Activité Physique Adaptée - CDOS Savoie, Chambéry
  - CH Chambéry, Chambéry
  - Activité Physique Adaptée - DAHLIR 63, Clermont-Ferrand
  - CHU Clermont-Ferrand - ONCOLOGIE, Clermont-Ferrand
  - CHU Clermont-Ferrand - Urologie, Clermont-Ferrand
  - Activité Physique Adaptée - CDOS Isère, Grenoble
  - CHU Grenoble - Urologie, Grenoble
  - Activité Physique Adaptée - DAHLIR 43, Le Puy-en-Velay
  - CH Le Puy en Velay, Le Puy-en-Velay
  - HCL - Hôpital Edouard Herriot, Lyon
  - HCL - Hôpital Croix Rousse, Lyon
  - Activité Physique Adaptée - DAHLIR 69, Lyon
  - CLB - Oncologie, Lyon
  - CLB - Radiothérapie, Lyon
  - HCL - CH Lyon Sud, Lyon
  - Activité Physique Adaptée - CDOS Ardèche, Privas
  - CH Roanne, Roanne
  - Activité Physique Adaptée - DAPAP 42, Saint-Etienne
  - CHU Saint-Etienne - Oncologie, Saint-Etienne
  - CHU Saint-Etienne - Radiothérapie, Saint-Etienne
  - Hôpital Privé de la Loire, Saint-Etienne
  - Clinique du parc, Saint-Priest-en-Jarez
  - Activité Physique Adaptée - CDOS Drôme, Valence
  - Hôpitaux Drôme Nord - Valence, Valence
  - Radiologie Drôme-Ardèche - Valence, Valence

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bonn SE, Sjolander A, Lagerros YT, Wiklund F, Stattin P, Holmberg E, Gronberg H, Balter K. Physical activity and survival among men diagnosed with prostate cancer. Cancer Epidemiol Biomarkers Prev. 2015 Jan;24(1):57-64. doi: 10.1158/1055-9965.EPI-14-0707. Epub 2014 Dec 19. PMID 25527697
- [Background] Richman EL, Kenfield SA, Stampfer MJ, Paciorek A, Carroll PR, Chan JM. Physical activity after diagnosis and risk of prostate cancer progression: data from the cancer of the prostate strategic urologic research endeavor. Cancer Res. 2011 Jun 1;71(11):3889-95. doi: 10.1158/0008-5472.CAN-10-3932. Epub 2011 May 24. PMID 21610110
- [Background] Phillips SM, Stampfer MJ, Chan JM, Giovannucci EL, Kenfield SA. Physical activity, sedentary behavior, and health-related quality of life in prostate cancer survivors in the health professionals follow-up study. J Cancer Surviv. 2015 Sep;9(3):500-11. doi: 10.1007/s11764-015-0426-2. Epub 2015 Apr 16. PMID 25876555
- [Background] Steindorf K, Depenbusch J, Haussmann A, Tsiouris A, Schmidt L, Hermann S, Sieverding M, Wiskemann J, Ungar N. Change patterns and determinants of physical activity differ between breast, prostate, and colorectal cancer patients. Support Care Cancer. 2020 Jul;28(7):3207-3218. doi: 10.1007/s00520-019-05097-1. Epub 2019 Nov 13. PMID 31720802
- [Background] Blaney JM, Lowe-Strong A, Rankin-Watt J, Campbell A, Gracey JH. Cancer survivors' exercise barriers, facilitators and preferences in the context of fatigue, quality of life and physical activity participation: a questionnaire-survey. Psychooncology. 2013 Jan;22(1):186-94. doi: 10.1002/pon.2072. Epub 2011 Oct 6. PMID 23296635
- [Background] Livingston PM, Craike MJ, Salmon J, Courneya KS, Gaskin CJ, Fraser SF, Mohebbi M, Broadbent S, Botti M, Kent B; ENGAGE Uro-Oncology Clinicians' Group. Effects of a clinician referral and exercise program for men who have completed active treatment for prostate cancer: A multicenter cluster randomized controlled trial (ENGAGE). Cancer. 2015 Aug 1;121(15):2646-54. doi: 10.1002/cncr.29385. Epub 2015 Apr 15. PMID 25877784
- [Background] Tudor-Locke C, Lauzon N, Myers AM, Bell RC, Chan CB, McCargar L, Speechley M, Rodger NW. Effectiveness of the First step Program delivered by professionals versus peers. J Phys Act Health. 2009 Jul;6(4):456-62. doi: 10.1123/jpah.6.4.456. PMID 19842459
- [Background] Buman MP, Giacobbi PR Jr, Dzierzewski JM, Morgan AA, McCrae CS, Roberts BL, Marsiske M. Peer Volunteers Improve Long-Term Maintenance of Physical Activity With Older Adults: A Randomized Controlled Trial. J Phys Act Health. 2011 Sep;8(s2):S257-S266. doi: 10.1123/jpah.8.s2.s257. PMID 28829716
- [Background] Pinto BM, Stein K, Dunsiger S. Peers promoting physical activity among breast cancer survivors: A randomized controlled trial. Health Psychol. 2015 May;34(5):463-72. doi: 10.1037/hea0000120. Epub 2014 Aug 11. PMID 25110844
- [Background] Galvao DA, Newton RU, Girgis A, Lepore SJ, Stiller A, Mihalopoulos C, Gardiner RA, Taaffe DR, Occhipinti S, Chambers SK. Randomized controlled trial of a peer led multimodal intervention for men with prostate cancer to increase exercise participation. Psychooncology. 2018 Jan;27(1):199-207. doi: 10.1002/pon.4495. Epub 2017 Jul 27. PMID 28685892
- [Background] Baudot A, Barth N, Colas C, Garros M, Garcin A, Oriol M, Roche F, Chauvin F, Mottet N, Hupin D; on behalf the Acti-Pair investigators. The physical activity experience of prostate cancer patients: a multicentre peer motivation monitoring feasibility study. The Acti-Pair study. Pilot Feasibility Stud. 2022 Jan 21;8(1):12. doi: 10.1186/s40814-022-00966-9. PMID 35063040
- [Derived] Baudot A, Fayolle E, Garros M, Barth N, Colin F, Presles E, Oriol M, Collange F, Chauvin F, Bourmaud A, Hupin D. Impact of the Acti-Pair programme on physical activity in patients with prostate cancer: protocol of the Acti-Pair 2 stepped-wedge cluster randomised trial. BMJ Open Sport Exerc Med. 2024 Dec 22;10(4):e002344. doi: 10.1136/bmjsem-2024-002344. eCollection 2024. PMID 39717077